CLINICAL TRIAL: NCT02262598
Title: Bioequivalence of 40 mg Telmisartan / 12.5 mg HCTZ of Fixed Dose Combination Compared to Its Monocomponents in Healthy Male Volunteers (an Open-label, Randomised, Single-dose, Two-way Crossover Study)
Brief Title: Bioequivalence of Telmisartan / HCTZ of Fixed Dose Combination Compared to Its Monocomponents in Healthy Male Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Boehringer Ingelheim (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 502.437
Record Dates: First submitted 2014-10-09; First posted 2014-10-13 (Estimated); Last update posted 2014-10-13 (Estimated); Status verified 2014-10

CONDITIONS: Healthy
MeSH Terms: interventions — Telmisartan

ARMS (2):
- Telmisartan/HCTZ fixed dose (Experimental)
  Interventions: Drug: Telmisartan/HCTZ fixed dose
- Telmisartan and HCTZ monocomponents (Active Comparator)
  Interventions: Drug: Telmisartan; Drug: Hydrochlorthiazide (HCTZ)

INTERVENTIONS:
Drug: Telmisartan
  Arms: Telmisartan and HCTZ monocomponents
Drug: Hydrochlorthiazide (HCTZ)
  Arms: Telmisartan and HCTZ monocomponents
Drug: Telmisartan/HCTZ fixed dose
  Arms: Telmisartan/HCTZ fixed dose

SUMMARY:
To establish the bioequivalence of fixed dose combination of 40 mg telmisartan / 12.5 mg HCTZ vs. its monocomponents

ELIGIBILITY:
Inclusion Criteria:

1. Healthy males according to the following criteria:

   Based upon a complete medical history, the physical examination (physical findings and measurements of height and body weight), vital signs (blood pressure (BP), pulse rate (PR)), 12-lead ECG (electrocardiogram), clinical laboratory tests
   * No finding of clinical relevance
   * No evidence of a clinically relevant concomitant disease
2. Age ≥20 years and Age ≤35 years
3. BMI ≥ 17.6 kg/m2 and BMI ≤ 25.0 kg/m2 (Body Mass Index)
4. Signed and dated written informed consent prior to admission to the study in accordance with Good Clinical Practice (GCP)(MHW Ordinance No. 28, as of Mar. 27, 1997) and the local legislation.

Exclusion Criteria:

1. Gastrointestinal, hepatic, renal, respiratory, cardiovascular, metabolic, immunological or hormonal disorders
2. Surgery of gastrointestinal tract (except appendectomy)
3. Diseases of the central nervous system (such as epilepsy) or psychiatric disorders or neurological disorders
4. History of relevant orthostatic hypotension, fainting spells or blackouts.
5. Chronic or relevant acute infections
6. History of allergy/hypersensitivity (including drug allergy) which is deemed relevant to the trial as judged by the investigator
7. Positive result for Hepatitis B virus surface antigen (HBsAg), anti Hepatitis C virus (HCV) anti bodies, syphilitic test or Human immunodeficiency virus (HIV) test
8. Intake of drugs with a long half-life (≥24 hours) within at least one month or less than 10 half-lives of the respective drug prior to administration or during the trial
9. Use of drugs which might reasonably influence the results of the trial based on the knowledge at the time of protocol preparation within 10 days prior to administration or during the trial.
10. Participation in another trial with an investigational drug within four months prior to administration or during the trial
11. Smoker (more than 20 cigarettes/day)
12. Inability to refrain from smoking during hospitalisation
13. Alcohol abuse (more than 60 g/day as ethanol ex.) three middle sized bottles of beer / three gous (equivalent to 540 mL) of sake)
14. Drug abuse
15. Blood donation (more than 100 mL within four weeks prior to administration or during the trial)
16. Excessive physical activities (within one week prior to administration or during the trial)
17. Any laboratory value outside the reference range that is of clinical relevance
18. Inability to comply with dietary regimen of study centre
19. Any other volunteers whom, the principal investigator or sub investigator would not allow to participate this study

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-09; Primary Completion 2004-10 (Actual)

PRIMARY OUTCOMES:
AUC0-tz (area under the concentration-time curve of the analyte in plasma over the time interval from 0 to the last quantifiable data point) | Up to 72 hours after drug administration
Cmax (maximum measured concentration of the analyte in plasma) | Up to 72 hours after drug administration

SECONDARY OUTCOMES:
AUC0-∞ (area under the concentration-time curve of the analyte in plasma over the time interval from 0 extrapolated to infinity) | Up to 72 hours after drug administration
tmax (time from dosing to the maximum concentration of the analyte in plasma) | Up to 72 hours after drug administration
λz (terminal rate constant of the analyte in plasma) | Up to 72 hours after drug administration
t1/2 (terminal half-life of the analyte in plasma) | Up to 72 hours after drug administration
MRTpo (mean residence time of the analyte in the body after po administration) | Up to 72 hours after drug administration
Number of participants with abnormal findings in physical examination | Up to 9 days after last drug administration
Number of participants with clinically significant findings in vital signs | Up to 9 days after last drug administration
Number of participants with clinically significant findings in 12-lead ECG (electrocardiogram) | Up to 9 days after last drug administration
Number of participants with clinically significant findings in laboratory parameters | Up to 9 days after last drug administration
Number of participants with adverse events | Up to 9 days after last drug administration